CLINICAL TRIAL: NCT03926741
Title: Methods to Identify and Treat Severe Asthma Patients Project 1: GSNOR Phenotyping and GSNO Challenge
Brief Title: GSNOR Phenotyping/GSNO Challenge in Severe Asthma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: James Reynolds (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Case Western Reserve University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, James Reynolds, Professor of Anesthesiology & Perioperative Medicine, Case Western Reserve University
Organization: Case Western Reserve University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-17-11; 5P01HL158507 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-04-24 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Asthma; Healthy Volunteers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GSNOR Challenge testing (Experimental): patient will use a nebulizer to inhale (breathe in) a solution of GSNO followed by repeated measurements of airway function (breathing tests)
  Interventions: Drug: GSNO

INTERVENTIONS:
Drug: GSNO — patient will use a nebulizer to inhale (breathe in) a solution of GSNO followed by repeated measurements of airway function (breathing tests)

SUMMARY:
Asthma is caused by or worsened by different things in different people. It is because of these differences that not all people with asthma respond the same to all treatments and medicines. If the investigators can better identify the changes in the airways or breathing pipes in patients with asthma, the investigators may be able to help patients make better choices about the medicines or treatments that are most likely to work best for each patient.

This research study is about one specific factor that is known to affect asthma in some patients. It involves an increase in the activity of an enzyme that is in people's airways. An enzyme is something that helps a chemical reaction to occur. The enzyme the investigators are studying in this research study is called GSNOR (S-nitrosoglutathione reductase) , and when the activity of this enzyme is increased, the result is that there is less GSNO (S-nitrosoglutathione) . GSNO is a chemical that protects people's airways. The initials stand for S-nitrosoglutathione, (pronounced s-nahy-troh-soh-gloo-tuh-thahy-ohn), and it is naturally produced by the body. It has an important role in regulating respiratory function (breathing) and preventing inflammation (swelling) in the respiratory tract (throat, airways, and lungs).

The amount of GSNO found in the body is controlled by the enzyme GSNOR (S-nitrosoglutathione reductase). GSNOR breaks down GSNO. Too much GSNOR leads to low levels of GSNO, and that can cause inflammation (swelling) and loss of airway function in some asthma patients.

The only way to measure GSNOR levels currently is with a bronchoscopy procedure where a scope is inserted into the patient's airways, often under sedation. This research study is being done to test the accuracy of another type of test that can be done in the doctor's office, rather than in a procedure area. This non-invasive diagnostic test, called a GSNO Challenge test, may be able to identify which asthma patients have increased activity of the airway enzyme GSNOR. The investigators are also studying the phenotypes (observable traits) in asthma patients with increased levels of GSNOR. If this research study is successful, in the future (after this research study is done). The investigators may be able to offer a cost-effective and non-invasive way to identify patients who have higher GSNOR activity levels and offer personalized treatments.

The GSNO Challenge test includes giving an investigational drug to breathe in (inhale). The investigational drug is GSNO. "Investigational" means the drug is not approved by any regulatory agencies including the Food and Drug Administration (FDA), and is still being tested for safety and effectiveness. The research is registered with the FDA, but again the GSNO treatment in this study (administered during the GSNO challenge testing) is not an approved treatment or diagnostic test for asthma.

DETAILED DESCRIPTION:
S-nitrosylation signaling is relevant to a broad range of diseases, including severe asthma. Work in the Severe Asthma Research Program (SARP) and other research networks has established that asthma is remarkably heterogeneous. The response to standard asthmatic therapies is sub-optimal in many patients. Targeting expected responders, or personalizing approach to treatment, would lead to improved outcomes and decreased treatment costs. Furthermore, since patients with asthma that is not responsive to standard therapies are highly symptomatic despite standard therapy, this subset may derive particular benefit from a personalized approach that includes clinical phenotyping, directed diagnostic testing to confirm underlying pathophysiology, and treatment directed specifically towards those findings.

The classical conceptualization of asthma as a disease of allergic inflammation is based on findings that many patients with asthma have a "Th2 high" phenotype characterized by high circulating levels of IgE, eosinophils and periostin. Patients with these features are particularly amenable to exciting, new antibody-based therapies. However, many patients are not in this phenotype, and, within the generalized phenotype, there is a Gaussian distribution of response. Further, these antibody treatments tend to be expensive and require parenteral administration. A myriad of alternative potential targets has been identified in patients with asthma who do not respond to standard asthma therapies, ranging from high levels of airway chitinase to low levels of vitamin D.

Early work documenting the presence of S-nitrosothiols (SNOs) in human airways and characterizing the potent bronchodilator activity of S-nitrosoglutathione (GSNO) led us to consider that in some patients asthma may represent a disorder in pulmonary SNO homeostasis. The focus of this study is on the subset of patients with asthma who have increased airway S-nitrosoglutathione reductase (GSNOR) activity. Increased activity of GSNOR results in a reduction in the available GSNO, resulting in increased smooth muscle constriction, and increased inflammation. This is a highly targetable process for which specific therapeutic agents are now becoming available. This approach can provide a paradigm for other personalized strategies. Identifying alternative approaches for patients with asthma do not respond to standard asthma therapies has important public health implications. The investigators conservatively estimate that formulation of personalized asthma therapies, including the current study, could halve the morbidity and societal costs of asthma. This in turn would result in fewer disease-related deaths and billions of dollars in economic savings per year in the US - the current annual costs of asthma to the American economy are estimated at $56 billion.

Preliminary work from the Severe Asthma Research Program suggests that patients with increased GSNOR activity and increased catabolism of the endogenous bronchodilator GSNO17 have characteristic phenotypic features (younger age, earlier onset of asthma, higher IgE), but this work needs to be expanded through a combination of mechanistic assessments and clinical testing. The investigators have shown in preliminary work that GSNOR activity in bronchoalveolar lavage (BAL) fluid and in cell lysates from BAL fluid is higher on average in subjects with asthma compared with healthy volunteers. The investigators have further shown the relevance of this finding to asthma in that there is a relationship between GSNOR activity and airway hyper-responsiveness, a hallmark of asthma. The significant linear association between GSNOR activity and the concentration of methacholine that provokes a 20% fall in FEV1 (Forced Expiratory Volume in 1 Second) in subjects with asthma but not in healthy volunteers. While the investigators have shown that GSNOR activity is higher on average in subjects with asthma compared with healthy volunteers, activity levels are quite variable across the spectrum of asthma severity. Accurately identifying patients with asthma who have elevated GSNOR activity levels for targeted therapies is an essential next step.

In the preliminary data, GSNOR activity was measured directly using bronchoscopic techniques to collect BAL fluid and directly measure activity levels. While our experience in the Severe Asthma Research Program shows that bronchoscopies can be done safely in subjects with asthma, it will be important to develop non-invasive methodology to identify patients with asthma and elevated GSNOR activity in order to make if more practical and feasible to test and use targeted treatments. The purpose of this protocol is to confirm previous work demonstrating that subjects with asthma have higher GSNOR activity levels than healthy volunteers, expand our ability to predict who will have elevated GSNOR activity levels based on clinical phenotype, and to develop non-invasive and point of care testing that can accurately identify those with elevated GSNOR levels.

ELIGIBILITY:
Inclusion Criteria:

For subjects with Asthma

* Adult males or females age ≥ 18 and ≤ 50 years at the time of enrollment
* Non-smoker
* Physician diagnosis of asthma for at least one year
* FEV1 bronchodilator reversibility > 12% or methacholine PC20 < 16 mg/ml (historical methacholine data from previous NIH trials including SARP and AsthmaNet will be allowed)
* Baseline post maximal bronchodilator FEV1 >55% predicted

Healthy Volunteers

* Adult males or females age ≥ 18 and ≤ 50 years at time of enrollment
* Non-smoker
* No history of asthma, chronic obstructive pulmonary disease (COPD), or other chronic lung disease
* No history of severe allergic/atopic disease requiring immunotherapy or immunomodulators

Exclusion Criteria

-> 5 pack year smoking history

* Body mass index (BMI) > 45
* Unable to perform repeatable consistent efforts in pulmonary function testing
* Individuals with prior diagnosis of vocal cord dysfunction or an anatomic anomaly that would increase the risks associated with the bronchoscopy procedure
* Prior diagnosis of cystic fibrosis, COPD, or other additional lung disease that in the investigator's opinion would make participant unsuitable for study participation
* History of premature birth before 35 weeks gestation
* Planning to relocate away from the clinical center (Cleveland, Ohio or central Indiana) area before study completion
* Lack of reliable communications channel (hard-wire phone, cell phone, email for follow-up contacts after bronchoscopy)
* Allergic to anesthetic medication(s) that would prevent participation in the study's bronchoscopy
* Blood pressure parameters outside the normal range of 90-180 mm Hg systolic and 50-100 mm Hg diastolic at time of screening
* Individuals with diabetes mellitus (type 1 or type 2)
* Individuals with renal failure or creatinine > 1.8 mg/dl at time of screening
* Individuals who are pregnant, breastfeeding, or are unwilling to use a medically acceptable method of birth control (as indicated on the Birth Control Methods Reference Card) from the time of consent until the end of the study to avoid pregnancy
* Individuals who report additional chronic diseases requiring medication of the heart, lungs, kidney, liver, brain, etc., or afflicted with any acute or chronic pathology that in the opinion of the screening physician makes them unsuitable for study such as coronary artery disease
* Asthma exacerbation requiring oral corticosteroids within the previous 30 days (can be rescreened)
* More than 3 exacerbations within the past 6 months
* Intubated for asthma within the past 12 months
* Respiratory or other infection requiring systemic antibiotics within the previous 14 days (can be rescreened)
* Current use of a vitamin K antagonist (warfarin) or other anticoagulant (e.g., heparin, clopidogrel, enoxaparin or dalteparin)
* Current use of beta-adrenergic blockers, tricyclic antidepressants, meperidine (or related central nervous system (CNS) agents), or nitrates
* Unable or unwilling to withhold medications prior to certain study procedures (skin test, spirometry, methacholine challenge)
* Inherited or acquired blood coagulation disorder, congenital methemoglobinemia, or a familial hemoglobinopathy that impacts oxygen delivery (e.g., sickle cell)
* Any illness, condition or recent surgeries that may increase the risks associated with the study
* Participation in any investigational drug study other than the Airway pH Study within the 4 week period prior to screening.
* Any acute viral illness, including active COVID-19 infection or acute viral respiratory symptoms; can rescreen 4 weeks after positive test result.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Airway GSNOR comparison | Baseline
  Airway GSNOR will be compared among the two different groups (Asthma and Healthy Volunteers).
Airway GSNOR comparison | 3 months
  Airway GSNOR will be compared among the two different groups (Asthma and Healthy Volunteers).

SECONDARY OUTCOMES:
Fractional Exhaled Nitric Oxide (FeNO) levels changes | Baseline
  FeNO measurements will be compared among the two different groups (Asthma and Healthy Volunteers).
Fractional Exhaled Nitric Oxide (FeNO) levels changes | 3 months
  FeNO measurements will be compared among the two different groups (Asthma and Healthy Volunteers).

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Ross, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification and analysis will be shared.
Supporting Information: SAP, CSR
Time Frame: Available Immediately following publication. No end date
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Irie T, Sips PY, Kai S, Kida K, Ikeda K, Hirai S, Moazzami K, Jiramongkolchai P, Bloch DB, Doulias PT, Armoundas AA, Kaneki M, Ischiropoulos H, Kranias E, Bloch KD, Stamler JS, Ichinose F. S-Nitrosylation of Calcium-Handling Proteins in Cardiac Adrenergic Signaling and Hypertrophy. Circ Res. 2015 Oct 9;117(9):793-803. doi: 10.1161/CIRCRESAHA.115.307157. Epub 2015 Aug 10. PMID 26259881
- [Background] Dweik RA, Comhair SA, Gaston B, Thunnissen FB, Farver C, Thomassen MJ, Kavuru M, Hammel J, Abu-Soud HM, Erzurum SC. NO chemical events in the human airway during the immediate and late antigen-induced asthmatic response. Proc Natl Acad Sci U S A. 2001 Feb 27;98(5):2622-7. doi: 10.1073/pnas.051629498. Epub 2001 Feb 20. PMID 11226289
- [Background] Moore WC, Evans MD, Bleecker ER, Busse WW, Calhoun WJ, Castro M, Chung KF, Erzurum SC, Curran-Everett D, Dweik RA, Gaston B, Hew M, Israel E, Mayse ML, Pascual RM, Peters SP, Silveira L, Wenzel SE, Jarjour NN; National Heart, Lung, and Blood Institute's Severe Asthma Research Group. Safety of investigative bronchoscopy in the Severe Asthma Research Program. J Allergy Clin Immunol. 2011 Aug;128(2):328-336.e3. doi: 10.1016/j.jaci.2011.02.042. Epub 2011 Apr 15. PMID 21496892
- [Background] Auten RL, Mason SN, Whorton MH, Lampe WR, Foster WM, Goldberg RN, Li B, Stamler JS, Auten KM. Inhaled ethyl nitrite prevents hyperoxia-impaired postnatal alveolar development in newborn rats. Am J Respir Crit Care Med. 2007 Aug 1;176(3):291-9. doi: 10.1164/rccm.200605-662OC. Epub 2007 May 3. PMID 17478622
- [Background] Colagiovanni DB, Borkhataria D, Looker D, Schuler D, Bachmann C, Sagelsdorff P, Honarvar N, Rosenthal GJ. Preclinical 28-day inhalation toxicity assessment of s-nitrosoglutathione in beagle dogs and Wistar rats. Int J Toxicol. 2011 Oct;30(5):466-77. doi: 10.1177/1091581811412084. Epub 2011 Aug 25. PMID 21868767
- [Background] Foster MW, Hess DT, Stamler JS. Protein S-nitrosylation in health and disease: a current perspective. Trends Mol Med. 2009 Sep;15(9):391-404. doi: 10.1016/j.molmed.2009.06.007. Epub 2009 Aug 31. PMID 19726230
- [Background] Haldar SM, Stamler JS. S-nitrosylation: integrator of cardiovascular performance and oxygen delivery. J Clin Invest. 2013 Jan;123(1):101-10. doi: 10.1172/JCI62854. Epub 2013 Jan 2. PMID 23281416
- [Background] Marshall HE, Hess DT, Stamler JS. S-nitrosylation: physiological regulation of NF-kappaB. Proc Natl Acad Sci U S A. 2004 Jun 15;101(24):8841-2. doi: 10.1073/pnas.0403034101. Epub 2004 Jun 8. No abstract available. PMID 15187230
- [Background] Savidge TC, Urvil P, Oezguen N, Ali K, Choudhury A, Acharya V, Pinchuk I, Torres AG, English RD, Wiktorowicz JE, Loeffelholz M, Kumar R, Shi L, Nie W, Braun W, Herman B, Hausladen A, Feng H, Stamler JS, Pothoulakis C. Host S-nitrosylation inhibits clostridial small molecule-activated glucosylating toxins. Nat Med. 2011 Aug 21;17(9):1136-41. doi: 10.1038/nm.2405. PMID 21857653
- [Background] Prasad R, Giri S, Nath N, Singh I, Singh AK. GSNO attenuates EAE disease by S-nitrosylation-mediated modulation of endothelial-monocyte interactions. Glia. 2007 Jan 1;55(1):65-77. doi: 10.1002/glia.20436. PMID 17019693
- [Background] Savidge TC, Newman P, Pothoulakis C, Ruhl A, Neunlist M, Bourreille A, Hurst R, Sofroniew MV. Enteric glia regulate intestinal barrier function and inflammation via release of S-nitrosoglutathione. Gastroenterology. 2007 Apr;132(4):1344-58. doi: 10.1053/j.gastro.2007.01.051. Epub 2007 Feb 1. PMID 17408650
- [Background] Marshall HE, Potts EN, Kelleher ZT, Stamler JS, Foster WM, Auten RL. Protection from lipopolysaccharide-induced lung injury by augmentation of airway S-nitrosothiols. Am J Respir Crit Care Med. 2009 Jul 1;180(1):11-8. doi: 10.1164/rccm.200807-1186OC. Epub 2009 Mar 26. PMID 19324975
- [Background] Que LG, Liu L, Yan Y, Whitehead GS, Gavett SH, Schwartz DA, Stamler JS. Protection from experimental asthma by an endogenous bronchodilator. Science. 2005 Jun 10;308(5728):1618-21. doi: 10.1126/science.1108228. Epub 2005 May 26. PMID 15919956
- [Background] Snyder AH, McPherson ME, Hunt JF, Johnson M, Stamler JS, Gaston B. Acute effects of aerosolized S-nitrosoglutathione in cystic fibrosis. Am J Respir Crit Care Med. 2002 Apr 1;165(7):922-6. doi: 10.1164/ajrccm.165.7.2105032. PMID 11934715
- [Background] Jenkins KT. Nitrogen compounds. Hamilton & hardy's industrial toxicology. John Wiley & Sons, Inc.; 2015:363-370.
- [Background] Marozkina NV, Wang XQ, Stsiapura V, Fitzpatrick A, Carraro S, Hawkins GA, Bleecker E, Meyers D, Jarjour N, Fain SB, Wenzel S, Busse W, Castro M, Panettieri RA Jr, Moore W, Lewis SJ, Palmer LA, Altes T, de Lange EE, Erzurum S, Teague WG, Gaston B. Phenotype of asthmatics with increased airway S-nitrosoglutathione reductase activity. Eur Respir J. 2015 Jan;45(1):87-97. doi: 10.1183/09031936.00042414. Epub 2014 Oct 30. PMID 25359343
- [Background] Que LG, Yang Z, Stamler JS, Lugogo NL, Kraft M. S-nitrosoglutathione reductase: an important regulator in human asthma. Am J Respir Crit Care Med. 2009 Aug 1;180(3):226-31. doi: 10.1164/rccm.200901-0158OC. Epub 2009 Apr 24. PMID 19395503
- [Background] Wysocki K, Park SY, Bleecker E, Busse W, Castro M, Chung KF, Gaston B, Erzurum S, Israel E, Teague WG, Moore CG, Wenzel S. Characterization of factors associated with systemic corticosteroid use in severe asthma: data from the Severe Asthma Research Program. J Allergy Clin Immunol. 2014 Mar;133(3):915-8. doi: 10.1016/j.jaci.2013.10.031. Epub 2013 Dec 9. No abstract available. PMID 24332222
- [Background] Moore WC, Meyers DA, Wenzel SE, Teague WG, Li H, Li X, D'Agostino R Jr, Castro M, Curran-Everett D, Fitzpatrick AM, Gaston B, Jarjour NN, Sorkness R, Calhoun WJ, Chung KF, Comhair SA, Dweik RA, Israel E, Peters SP, Busse WW, Erzurum SC, Bleecker ER; National Heart, Lung, and Blood Institute's Severe Asthma Research Program. Identification of asthma phenotypes using cluster analysis in the Severe Asthma Research Program. Am J Respir Crit Care Med. 2010 Feb 15;181(4):315-23. doi: 10.1164/rccm.200906-0896OC. Epub 2009 Nov 5. PMID 19892860
- [Background] Chupp GL, Lee CG, Jarjour N, Shim YM, Holm CT, He S, Dziura JD, Reed J, Coyle AJ, Kiener P, Cullen M, Grandsaigne M, Dombret MC, Aubier M, Pretolani M, Elias JA. A chitinase-like protein in the lung and circulation of patients with severe asthma. N Engl J Med. 2007 Nov 15;357(20):2016-27. doi: 10.1056/NEJMoa073600. PMID 18003958
- [Background] Searing DA, Zhang Y, Murphy JR, Hauk PJ, Goleva E, Leung DY. Decreased serum vitamin D levels in children with asthma are associated with increased corticosteroid use. J Allergy Clin Immunol. 2010 May;125(5):995-1000. doi: 10.1016/j.jaci.2010.03.008. Epub 2010 Apr 9. PMID 20381849
- [Background] Ying S, O'Connor B, Ratoff J, Meng Q, Mallett K, Cousins D, Robinson D, Zhang G, Zhao J, Lee TH, Corrigan C. Thymic stromal lymphopoietin expression is increased in asthmatic airways and correlates with expression of Th2-attracting chemokines and disease severity. J Immunol. 2005 Jun 15;174(12):8183-90. doi: 10.4049/jimmunol.174.12.8183. PMID 15944327
- [Background] Bel EH, Wenzel SE, Thompson PJ, Prazma CM, Keene ON, Yancey SW, Ortega HG, Pavord ID; SIRIUS Investigators. Oral glucocorticoid-sparing effect of mepolizumab in eosinophilic asthma. N Engl J Med. 2014 Sep 25;371(13):1189-97. doi: 10.1056/NEJMoa1403291. Epub 2014 Sep 8. PMID 25199060
- [Background] Wenzel S, Ford L, Pearlman D, Spector S, Sher L, Skobieranda F, Wang L, Kirkesseli S, Rocklin R, Bock B, Hamilton J, Ming JE, Radin A, Stahl N, Yancopoulos GD, Graham N, Pirozzi G. Dupilumab in persistent asthma with elevated eosinophil levels. N Engl J Med. 2013 Jun 27;368(26):2455-66. doi: 10.1056/NEJMoa1304048. Epub 2013 May 21. PMID 23688323
- [Background] Busse WW, Morgan WJ, Gergen PJ, Mitchell HE, Gern JE, Liu AH, Gruchalla RS, Kattan M, Teach SJ, Pongracic JA, Chmiel JF, Steinbach SF, Calatroni A, Togias A, Thompson KM, Szefler SJ, Sorkness CA. Randomized trial of omalizumab (anti-IgE) for asthma in inner-city children. N Engl J Med. 2011 Mar 17;364(11):1005-15. doi: 10.1056/NEJMoa1009705. PMID 21410369
- [Background] Holgate ST. Trials and tribulations in identifying new biologic treatments for asthma. Trends Immunol. 2012 May;33(5):238-46. doi: 10.1016/j.it.2012.02.003. Epub 2012 Mar 20. PMID 22436378
- [Background] Barnes PJ. Severe asthma: advances in current management and future therapy. J Allergy Clin Immunol. 2012 Jan;129(1):48-59. doi: 10.1016/j.jaci.2011.11.006. PMID 22196524
- [Background] Comhair SA, Erzurum SC. Redox control of asthma: molecular mechanisms and therapeutic opportunities. Antioxid Redox Signal. 2010 Jan;12(1):93-124. doi: 10.1089/ars.2008.2425. PMID 19634987
- [Background] Sun X, Qiu J, Strong SA, Green LS, Wasley JW, Colagiovanni DB, Mutka SC, Blonder JP, Stout AM, Richards JP, Chun L, Rosenthal GJ. Structure-activity relationships of pyrrole based S-nitrosoglutathione reductase inhibitors: pyrrole regioisomers and propionic acid replacement. Bioorg Med Chem Lett. 2011 Jun 15;21(12):3671-5. doi: 10.1016/j.bmcl.2011.04.086. Epub 2011 Apr 24. PMID 21570838
- [Background] Sun X, Wasley JW, Qiu J, Blonder JP, Stout AM, Green LS, Strong SA, Colagiovanni DB, Richards JP, Mutka SC, Chun L, Rosenthal GJ. Discovery of s-nitrosoglutathione reductase inhibitors: potential agents for the treatment of asthma and other inflammatory diseases. ACS Med Chem Lett. 2011 Mar 11;2(5):402-6. doi: 10.1021/ml200045s. eCollection 2011 May 12. PMID 24900320
- [Background] Winer RA, Qin X, Harrington T, Moorman J, Zahran H. Asthma incidence among children and adults: findings from the Behavioral Risk Factor Surveillance system asthma call-back survey--United States, 2006-2008. J Asthma. 2012 Feb;49(1):16-22. doi: 10.3109/02770903.2011.637594. PMID 22236442
- [Background] Bryan NS, Bian K, Murad F. Discovery of the nitric oxide signaling pathway and targets for drug development. Front Biosci (Landmark Ed). 2009 Jan 1;14(1):1-18. doi: 10.2741/3228. PMID 19273051
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Lima B, Forrester MT, Hess DT, Stamler JS. S-nitrosylation in cardiovascular signaling. Circ Res. 2010 Mar 5;106(4):633-46. doi: 10.1161/CIRCRESAHA.109.207381. PMID 20203313
- [Background] Hess DT, Foster MW, Stamler JS. Assays for S-nitrosothiols and S-nitrosylated proteins and mechanistic insights into cardioprotection. Circulation. 2009 Jul 21;120(3):190-3. doi: 10.1161/CIRCULATIONAHA.109.876607. Epub 2009 Jul 6. No abstract available. PMID 19581490
- [Background] Singh SP, Wishnok JS, Keshive M, Deen WM, Tannenbaum SR. The chemistry of the S-nitrosoglutathione/glutathione system. Proc Natl Acad Sci U S A. 1996 Dec 10;93(25):14428-33. doi: 10.1073/pnas.93.25.14428. PMID 8962068
- [Background] Schroeder RA, Cai C, Kuo PC. Endotoxin-mediated nitric oxide synthesis inhibits IL-1beta gene transcription in ANA-1 murine macrophages. Am J Physiol. 1999 Sep;277(3):C523-30. doi: 10.1152/ajpcell.1999.277.3.C523. PMID 10484338
- [Background] Xiong H, Zhu C, Li F, Hegazi R, He K, Babyatsky M, Bauer AJ, Plevy SE. Inhibition of interleukin-12 p40 transcription and NF-kappaB activation by nitric oxide in murine macrophages and dendritic cells. J Biol Chem. 2004 Mar 12;279(11):10776-83. doi: 10.1074/jbc.M313416200. Epub 2003 Dec 16. PMID 14679201
- [Background] Into T, Inomata M, Nakashima M, Shibata K, Hacker H, Matsushita K. Regulation of MyD88-dependent signaling events by S nitrosylation retards toll-like receptor signal transduction and initiation of acute-phase immune responses. Mol Cell Biol. 2008 Feb;28(4):1338-47. doi: 10.1128/MCB.01412-07. Epub 2007 Dec 17. PMID 18086890
- [Background] del Fresno C, Gomez-Garcia L, Caveda L, Escoll P, Arnalich F, Zamora R, Lopez-Collazo E. Nitric oxide activates the expression of IRAK-M via the release of TNF-alpha in human monocytes. Nitric Oxide. 2004 Jun;10(4):213-20. doi: 10.1016/j.niox.2004.04.007. PMID 15275867
- [Background] Gonzalez-Leon MC, Soares-Schanoski A, del Fresno C, Cimadevila A, Gomez-Pina V, Mendoza-Barbera E, Garcia F, Marin E, Arnalich F, Fuentes-Prior P, Lopez-Collazo E. Nitric oxide induces SOCS-1 expression in human monocytes in a TNF-alpha-dependent manner. J Endotoxin Res. 2006;12(5):296-306. doi: 10.1179/096805106X118843. PMID 17059693
- [Background] Marshall HE, Stamler JS. Inhibition of NF-kappa B by S-nitrosylation. Biochemistry. 2001 Feb 13;40(6):1688-93. doi: 10.1021/bi002239y. PMID 11327828
- [Background] Kelleher ZT, Matsumoto A, Stamler JS, Marshall HE. NOS2 regulation of NF-kappaB by S-nitrosylation of p65. J Biol Chem. 2007 Oct 19;282(42):30667-72. doi: 10.1074/jbc.M705929200. Epub 2007 Aug 24. PMID 17720813
- [Background] Gaston B, Reilly J, Drazen JM, Fackler J, Ramdev P, Arnelle D, Mullins ME, Sugarbaker DJ, Chee C, Singel DJ, Loscalzo J, Stamler JS. Endogenous nitrogen oxides and bronchodilator S-nitrosothiols in human airways. Proc Natl Acad Sci U S A. 1993 Dec 1;90(23):10957-61. doi: 10.1073/pnas.90.23.10957. PMID 8248198
- [Background] Liu L, Hausladen A, Zeng M, Que L, Heitman J, Stamler JS. A metabolic enzyme for S-nitrosothiol conserved from bacteria to humans. Nature. 2001 Mar 22;410(6827):490-4. doi: 10.1038/35068596. PMID 11260719
- [Background] Wei W, Li B, Hanes MA, Kakar S, Chen X, Liu L. S-nitrosylation from GSNOR deficiency impairs DNA repair and promotes hepatocarcinogenesis. Sci Transl Med. 2010 Feb 17;2(19):19ra13. doi: 10.1126/scitranslmed.3000328. PMID 20371487
- [Background] Crosswhite P, Sun Z. Nitric oxide, oxidative stress and inflammation in pulmonary arterial hypertension. J Hypertens. 2010 Feb;28(2):201-12. doi: 10.1097/HJH.0b013e328332bcdb. PMID 20051913
- [Background] Marozkina NV, Yemen S, Borowitz M, Liu L, Plapp M, Sun F, Islam R, Erdmann-Gilmore P, Townsend RR, Lichti CF, Mantri S, Clapp PW, Randell SH, Gaston B, Zaman K. Hsp 70/Hsp 90 organizing protein as a nitrosylation target in cystic fibrosis therapy. Proc Natl Acad Sci U S A. 2010 Jun 22;107(25):11393-8. doi: 10.1073/pnas.0909128107. Epub 2010 Jun 8. PMID 20534503
- [Background] Gaston B, Sears S, Woods J, Hunt J, Ponaman M, McMahon T, Stamler JS. Bronchodilator S-nitrosothiol deficiency in asthmatic respiratory failure. Lancet. 1998 May 2;351(9112):1317-9. doi: 10.1016/S0140-6736(97)07485-0. PMID 9643794
- [Background] Whalen EJ, Foster MW, Matsumoto A, Ozawa K, Violin JD, Que LG, Nelson CD, Benhar M, Keys JR, Rockman HA, Koch WJ, Daaka Y, Lefkowitz RJ, Stamler JS. Regulation of beta-adrenergic receptor signaling by S-nitrosylation of G-protein-coupled receptor kinase 2. Cell. 2007 May 4;129(3):511-22. doi: 10.1016/j.cell.2007.02.046. PMID 17482545
- [Background] Gaston B, Drazen JM, Loscalzo J, Stamler JS. The biology of nitrogen oxides in the airways. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):538-51. doi: 10.1164/ajrccm.149.2.7508323.
- [Background] Moya MP, Gow AJ, McMahon TJ, Toone EJ, Cheifetz IM, Goldberg RN, Stamler JS. S-nitrosothiol repletion by an inhaled gas regulates pulmonary function. Proc Natl Acad Sci U S A. 2001 May 8;98(10):5792-7. doi: 10.1073/pnas.091109498. Epub 2001 Apr 24. PMID 11320213
- [Background] McMahon TJ, Ahearn GS, Moya MP, Gow AJ, Huang YC, Luchsinger BP, Nudelman R, Yan Y, Krichman AD, Bashore TM, Califf RM, Singel DJ, Piantadosi CA, Tapson VF, Stamler JS. A nitric oxide processing defect of red blood cells created by hypoxia: deficiency of S-nitrosohemoglobin in pulmonary hypertension. Proc Natl Acad Sci U S A. 2005 Oct 11;102(41):14801-6. doi: 10.1073/pnas.0506957102. Epub 2005 Oct 3. PMID 16203976
- [Background] Moya MP, Gow AJ, Califf RM, Goldberg RN, Stamler JS. Inhaled ethyl nitrite gas for persistent pulmonary hypertension of the newborn. Lancet. 2002 Jul 13;360(9327):141-3. doi: 10.1016/S0140-6736(02)09385-6. PMID 12126827
- [Background] Green LS, Chun LE, Patton AK, Sun X, Rosenthal GJ, Richards JP. Mechanism of inhibition for N6022, a first-in-class drug targeting S-nitrosoglutathione reductase. Biochemistry. 2012 Mar 13;51(10):2157-68. doi: 10.1021/bi201785u. Epub 2012 Feb 28. PMID 22335564
- [Background] Colagiovanni DB, Drolet DW, Langlois-Forget E, Piche MP, Looker D, Rosenthal GJ. A nonclinical safety and pharmacokinetic evaluation of N6022: a first-in-class S-nitrosoglutathione reductase inhibitor for the treatment of asthma. Regul Toxicol Pharmacol. 2012 Feb;62(1):115-24. doi: 10.1016/j.yrtph.2011.12.012. Epub 2011 Dec 24. PMID 22210450
- [Background] Tan S, Hall IP, Dewar J, Dow E, Lipworth B. Association between beta 2-adrenoceptor polymorphism and susceptibility to bronchodilator desensitisation in moderately severe stable asthmatics. Lancet. 1997 Oct 4;350(9083):995-9. doi: 10.1016/S0140-6736(97)03211-X. PMID 9329515
- [Background] Israel E, Drazen JM, Liggett SB, Boushey HA, Cherniack RM, Chinchilli VM, Cooper DM, Fahy JV, Fish JE, Ford JG, Kraft M, Kunselman S, Lazarus SC, Lemanske RF, Martin RJ, McLean DE, Peters SP, Silverman EK, Sorkness CA, Szefler SJ, Weiss ST, Yandava CN. The effect of polymorphisms of the beta(2)-adrenergic receptor on the response to regular use of albuterol in asthma. Am J Respir Crit Care Med. 2000 Jul;162(1):75-80. doi: 10.1164/ajrccm.162.1.9907092. PMID 10903223
- [Background] Wechsler ME, Kunselman SJ, Chinchilli VM, Bleecker E, Boushey HA, Calhoun WJ, Ameredes BT, Castro M, Craig TJ, Denlinger L, Fahy JV, Jarjour N, Kazani S, Kim S, Kraft M, Lazarus SC, Lemanske RF Jr, Markezich A, Martin RJ, Permaul P, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Walter MJ, Wasserman SI, Israel E; National Heart, Lung and Blood Institute's Asthma Clinical Research Network. Effect of beta2-adrenergic receptor polymorphism on response to longacting beta2 agonist in asthma (LARGE trial): a genotype-stratified, randomised, placebo-controlled, crossover trial. Lancet. 2009 Nov 21;374(9703):1754-64. doi: 10.1016/S0140-6736(09)61492-6. PMID 19932356
- [Background] Martinez FD, Graves PE, Baldini M, Solomon S, Erickson R. Association between genetic polymorphisms of the beta2-adrenoceptor and response to albuterol in children with and without a history of wheezing. J Clin Invest. 1997 Dec 15;100(12):3184-8. doi: 10.1172/JCI119874. PMID 9399966
- [Background] Choudhry S, Que LG, Yang Z, Liu L, Eng C, Kim SO, Kumar G, Thyne S, Chapela R, Rodriguez-Santana JR, Rodriguez-Cintron W, Avila PC, Stamler JS, Burchard EG. GSNO reductase and beta2-adrenergic receptor gene-gene interaction: bronchodilator responsiveness to albuterol. Pharmacogenet Genomics. 2010 Jun;20(6):351-8. doi: 10.1097/FPC.0b013e328337f992. PMID 20335826
- [Background] Wu H, Romieu I, Sienra-Monge JJ, Estela Del Rio-Navarro B, Anderson DM, Jenchura CA, Li H, Ramirez-Aguilar M, Del Carmen Lara-Sanchez I, London SJ. Genetic variation in S-nitrosoglutathione reductase (GSNOR) and childhood asthma. J Allergy Clin Immunol. 2007 Aug;120(2):322-8. doi: 10.1016/j.jaci.2007.04.022. Epub 2007 Jun 1. PMID 17543375
- [Background] Moore PE, Ryckman KK, Williams SM, Patel N, Summar ML, Sheller JR. Genetic variants of GSNOR and ADRB2 influence response to albuterol in African-American children with severe asthma. Pediatr Pulmonol. 2009 Jul;44(7):649-54. doi: 10.1002/ppul.21033. PMID 19514054
- [Background] Kupczyk M, Wenzel S. U.S. and European severe asthma cohorts: what can they teach us about severe asthma? J Intern Med. 2012 Aug;272(2):121-32. doi: 10.1111/j.1365-2796.2012.02558.x. PMID 22630041
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Hess DT, Matsumoto A, Kim SO, Marshall HE, Stamler JS. Protein S-nitrosylation: purview and parameters. Nat Rev Mol Cell Biol. 2005 Feb;6(2):150-66. doi: 10.1038/nrm1569. PMID 15688001
- [Background] Seth D, Stamler JS. The SNO-proteome: causation and classifications. Curr Opin Chem Biol. 2011 Feb;15(1):129-36. doi: 10.1016/j.cbpa.2010.10.012. Epub 2010 Nov 17. PMID 21087893
- [Background] Haldar SM, Stamler JS. S-Nitrosylation at the interface of autophagy and disease. Mol Cell. 2011 Jul 8;43(1):1-3. doi: 10.1016/j.molcel.2011.06.014. PMID 21726803
- [Background] Asano K, Chee CB, Gaston B, Lilly CM, Gerard C, Drazen JM, Stamler JS. Constitutive and inducible nitric oxide synthase gene expression, regulation, and activity in human lung epithelial cells. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):10089-93. doi: 10.1073/pnas.91.21.10089. PMID 7524082
- [Background] Forrester MT, Thompson JW, Foster MW, Nogueira L, Moseley MA, Stamler JS. Proteomic analysis of S-nitrosylation and denitrosylation by resin-assisted capture. Nat Biotechnol. 2009 Jun;27(6):557-9. doi: 10.1038/nbt.1545. Epub 2009 May 31. PMID 19483679
- [Background] Yick CY, Zwinderman AH, Kunst PW, Grunberg K, Mauad T, Dijkhuis A, Bel EH, Baas F, Lutter R, Sterk PJ. Transcriptome sequencing (RNA-Seq) of human endobronchial biopsies: asthma versus controls. Eur Respir J. 2013 Sep;42(3):662-70. doi: 10.1183/09031936.00115412. Epub 2013 Jan 11. PMID 23314903
- [Background] Brown-Steinke K, deRonde K, Yemen S, Palmer LA. Gender differences in S-nitrosoglutathione reductase activity in the lung. PLoS One. 2010 Nov 16;5(11):e14007. doi: 10.1371/journal.pone.0014007. PMID 21103380
- [Background] Olson N, Kasahara DI, Hristova M, Bernstein R, Janssen-Heininger Y, van der Vliet A. Modulation of NF-kappaB and hypoxia-inducible factor--1 by S-nitrosoglutathione does not alter allergic airway inflammation in mice. Am J Respir Cell Mol Biol. 2011 Jun;44(6):813-23. doi: 10.1165/rcmb.2010-0035OC. Epub 2010 Aug 6. PMID 20693401
- [Background] Foster MW, Yang Z, Gooden DM, Thompson JW, Ball CH, Turner ME, Hou Y, Pi J, Moseley MA, Que LG. Proteomic characterization of the cellular response to nitrosative stress mediated by s-nitrosoglutathione reductase inhibition. J Proteome Res. 2012 Apr 6;11(4):2480-91. doi: 10.1021/pr201180m. Epub 2012 Mar 19. PMID 22390303
- [Background] COMROE JH Jr, FOWLER WS. Lung function studies. VI. Detection of uneven alveolar ventilation during a single breath of oxygen. Am J Med. 1951 Apr;10(4):408-13. doi: 10.1016/0002-9343(51)90285-9. No abstract available. PMID 14819046
- [Background] Greenwald R, Fitzpatrick AM, Gaston B, Marozkina NV, Erzurum S, Teague WG. Breath formate is a marker of airway S-nitrosothiol depletion in severe asthma. PLoS One. 2010 Jul 30;5(7):e11919. doi: 10.1371/journal.pone.0011919. PMID 20689836
- [Background] Schuler M, Faller H, Wittmann M, Schultz K. Asthma Control Test and Asthma Control Questionnaire: factorial validity, reliability and correspondence in assessing status and change in asthma control. J Asthma. 2016;53(4):438-45. doi: 10.3109/02770903.2015.1101134. Epub 2016 Jan 21. PMID 26539757
- [Background] Sullivan PW, Globe G, Ghushchyan VH, Campbell JD, Bender B, Magid DJ. Exploring asthma control cutoffs and economic outcomes using the Asthma Control Questionnaire. Ann Allergy Asthma Immunol. 2016 Sep;117(3):251-257.e2. doi: 10.1016/j.anai.2016.07.020. PMID 27613458
- [Background] Bateman ED, Esser D, Chirila C, Fernandez M, Fowler A, Moroni-Zentgraf P, FitzGerald JM. Magnitude of effect of asthma treatments on Asthma Quality of Life Questionnaire and Asthma Control Questionnaire scores: Systematic review and network meta-analysis. J Allergy Clin Immunol. 2015 Oct;136(4):914-22. doi: 10.1016/j.jaci.2015.03.023. Epub 2015 May 1. PMID 25936565
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Halldin CN, Doney BC, Hnizdo E. Changes in prevalence of chronic obstructive pulmonary disease and asthma in the US population and associated risk factors. Chron Respir Dis. 2015 Feb;12(1):47-60. doi: 10.1177/1479972314562409. Epub 2014 Dec 24. PMID 25540134
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836